CLINICAL TRIAL: NCT06719115
Title: A Randomized, Triple-blind, Placebo Controlled, Parallel Clinical Trial to Investigate the Safety and Efficacy of D-Mannose on Symptoms of Urinary Tract Infection in Women
Brief Title: A Clinical Trial to Investigate the Safety and Efficacy of D-Mannose on Symptoms of Urinary Tract Infection in Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: KEB Nutraceuticals USA, Inc. (Industry)
Collaborators: KGK Science Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 22KBCFD01
Record Dates: First submitted 2024-12-02; First posted 2024-12-05 (Actual); Last update posted 2024-12-05 (Actual); Status verified 2024-12

CONDITIONS: Urinary Tract Infection(UTI)
Keywords: Uncomplicated urinary tract infection
MeSH Terms: conditions — Urinary Tract Infections

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- UClear (Experimental): UClear contains 1.5g of D-Mannose. Participants will be instructed to take one dose twice a day for three days with or without food, starting on Day 1 (baseline visit). The product should be completely dissolved in a full glass of water and participants are instructed to take one dose in the morning and one dose in the afternoon. If a dose was missed participants were instructed to take the missed dose as soon as they remembered. Participants were advised not to exceed two doses daily.
  Interventions: Dietary Supplement: UClear
- Placebo (Placebo Comparator): Participants will be instructed to take one dose twice a day for three days with or without food, starting on Day 1 (baseline visit).The product should be completely dissolved in a full glass of water and participants are instructed to take one dose in the morning and one dose in the afternoon. If a dose was missed participants were instructed to take the missed dose as soon as they remembered. Participants were advised not to exceed two doses daily.
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: UClear — Take one dose twice a day for three days with or without food, starting on Day 1 (baseline visit).
  Arms: UClear
Other: Placebo — Take one dose twice a day for three days with or without food, starting on Day 1 (baseline visit).
  Arms: Placebo

SUMMARY:
The objective of this acute study was to investigate the safety and efficacy of UClear for the resolution of urinary tract infection (UTI) symptoms in women. The main questions it aims to answer is:

1. Is there a difference in proportion of participants with complete resolution of UTI symptoms at Day 4 between UClear and placebo
2. Is there a difference in change from baseline (Day 1) at Day 4 between UClear and placebo in Urinary Tract Infection Symptom Assessment (UTISA) symptom severity scores.

Participants will take UClear or placebo twice a day for 3 days with or without food, have 4 in clinical visits, and will be instructed to complete a quality of life (QoL) questionnaire during each visit and a UTISA questionnaire at follow-up (Day 7).

ELIGIBILITY:
Inclusion Criteria:

* Females between 18 and 75 years of age, inclusive, at screening
* Individuals not of child-bearing potential, defined as those who have undergone a sterilization procedure (e.g. hysterectomy, bilateral oophorectomy, bilateral tubal ligation, complete endometrial ablation) or have been post-menopausal for at least 1 year prior to screening Or,

Individuals of child-bearing potential must have a negative baseline urine pregnancy test and agree to use a medically approved method of birth control for the duration of the study. All hormonal birth control must have been in use for a minimum of three months. Acceptable methods of birth control include:

* Hormonal contraceptives including oral contraceptives, hormone birth control patch (Ortho Evra), vaginal contraceptive ring (NuvaRing), injectable contraceptives (Depo-Provera, Lunelle), or hormone implant (Norplant System)
* Double-barrier method
* Intrauterine devices
* Non-heterosexual lifestyle or agrees to use contraception if planning on changing to heterosexual partner(s)
* Vasectomy of partner at least 6 months prior to screening

  * At least two uncomplicated UTI symptoms defined by frequent, urgent, and painful urination, incomplete voiding, pelvic and low back pain, and blood in urine, as assessed by UTISA questionnaire
  * Positive urine dip stick test for nitrites or leukocytes
  * Agree to keep lifestyle, including dietary habits, physical activity patterns, and medications/supplements, consistent for the duration of the trial
  * Provided voluntary, written, informed consent to participate in the study

Exclusion Criteria:

* Individuals who are pregnant, breast feeding, or planning to become pregnant during the study
* Allergy, sensitivity, or intolerance to the investigational product, placebo, or rescue medication ingredients
* Clinical signs and symptoms of an upper UTI (ex. costovertebral pain or tenderness, nausea, vomiting, fever), as assessed by the QI
* Anatomical or functional urinary tract abnormalities and/or diagnosis of kidney or other urinary tract diseases/conditions, such as painful bladder syndrome, neurogenic bladder, and polycystic kidney disease, as assessed by the QI
* History of or current urological cancers
* Current use of an indwelling catheter or intermittent catheterization
* Type I or Type II diabetes
* Unstable hypertension. Treatment on a stable dose of medication for at least three months will be considered by the QI
* Self-reported confirmation of current or pre-existing thyroid condition. Treatment on a stable dose of medication for at least three months will be considered by the QI
* Self-reported confirmation of blood/bleeding disorders
* Individuals with an autoimmune disease or are immune compromised, as assessed by the QI
* Unstable metabolic disease or chronic diseases as assessed by the QI
* Current or history of any significant diseases of the gastrointestinal tract, as assessed by the QI
* History of or current diagnosis of liver diseases as assessed by the QI
* Participants who are within three days of the end of their menstruation, menstruating, or anticipating menstruation during the study
* Major surgery in the past three months or individuals who have planned surgery during the course of the study. Participants with minor surgery will be considered on a case-by-case basis by the QI
* Current use of prescribed medications, over-the-counter (OTC) medications, or supplements, food/ drinks which may affect the efficacy and/or safety of the IP (see Sections 12.4.6 and 12.4.7)
* Use of medical cannabinoid products
* Use of cannabinoid products and is unwilling to stop use for the duration of the study
* Alcohol intake average of >2 standard drinks per day as assessed by the QI
* Alcohol or drug abuse within the last 12 months
* Blood donation 30 days prior to baseline, during the study, or a planned donation within 30 days of the last study visit
* Participation in other clinical research studies 30 days prior to baseline, as assessed by the QI
* Individuals who are unable to give informed consent
* Any other condition or lifestyle factor, that, in the opinion of the QI, may adversely affect the participant's ability to complete the study or its measures or pose significant risk to the participant

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Actual)
Dates: Start 2023-05-03 (Actual); Primary Completion 2024-06-20 (Actual); Study Completion 2024-06-20 (Actual)

PRIMARY OUTCOMES:
The difference in proportion of participants with complete resolution of UTI symptoms at Day 4 between D-mannose and placebo | Day 1 to 4
  The difference in proportion of participants with complete resolution of UTI symptoms at Day 4 between D-mannose and placebo as defined as 0 points on all UTISA questionnaire components.
The difference in change between D-mannose and placebo in UTISA symptom severity scores | Day 1 to 4
  The difference in change from baseline (Day 1) at Day 4 between D-mannose and placebo in the frequency of urination
The difference in change between D-mannose and placebo in UTISA symptom severity scores | Day 1 to 4
  The difference in change from baseline (Day 1) at Day 4 between D-mannose and placebo in urgency of urination
The difference in change between D-mannose and placebo in UTISA symptom severity scores | Day 1 to 4
  The difference in change from baseline (Day 1) at Day 4 between D-mannose and placebo in painful/burning urination
The difference in change between D-mannose and placebo in UTISA symptom severity scores | Day 1 to 4
  The difference in change from baseline (Day 1) at Day 4 between D-mannose and placebo in incomplete voiding
The difference in change between D-mannose and placebo in UTISA symptom severity scores | Day 1 to 4
  The difference in change from baseline (Day 1) at Day 4 between D-mannose and placebo in pelvic pain
The difference in change between D-mannose and placebo in UTISA symptom severity scores | Day 1 to 4
  The difference in change from baseline (Day 1) at Day 4 between D-mannose and placebo in blood in urine

SECONDARY OUTCOMES:
The difference in proportion of participants with complete resolution of UTI symptoms between D-mannose and placebo | Day 1 to 2
  The difference in proportion of participants with complete resolution of UTI symptoms between D-mannose and placebo at Day 2
The difference in proportion of participants with complete resolution of UTI symptoms between D-mannose and placebo | Day 1 to 3
  The difference in proportion of participants with complete resolution of UTI symptoms between D-mannose and placebo at Day 3
The difference in the change in symptom severity scores from baseline between D-mannose and placebo | Day 1 to 2
  The difference in the change in symptom severity scores from baseline between D-mannose and placebo as assessed by UTISA questionnaire at Day 2
The difference in the change in symptom severity scores from baseline between D-mannose and placebo | Day 1 to 3
  The difference in the change in symptom severity scores from baseline between D-mannose and placebo as assessed by UTISA questionnaire at Day 3
The difference in the change in UTISA bother scores from baseline between D-mannose and placebo | Day 1 to 2
  The difference in the change in UTISA bother scores from baseline between D-mannose and placebo as assessed by UTISA questionnaire at Day 2
The difference in the change in UTISA bother scores from baseline between D-mannose and placebo | Day 1 to 3
  The difference in the change in UTISA bother scores from baseline between D-mannose and placebo as assessed by UTISA questionnaire at Day 3
The difference in the change in UTISA bother scores from baseline between D-mannose and placebo | Day 1 to 4
  The difference in the change in UTISA bother scores from baseline between D-mannose and placebo as assessed by UTISA questionnaire at Day 4
The difference in change in urine culture (multiple bacterial strains) from baseline between D-mannose and placebo | Day 1 to 2
  The difference in change in urine culture (multiple bacterial strains) from baseline between D-mannose and placebo at Day 2
The difference in change in urine culture (multiple bacterial strains) from baseline between D-mannose and placebo | Day 1 to 3
  The difference in change in urine culture (multiple bacterial strains) from baseline between D-mannose and placebo at Day 3
The difference in change in urine culture (multiple bacterial strains) from baseline between D-mannose and placebo | Day 1 to 4
  The difference in change in urine culture (multiple bacterial strains) from baseline between D-mannose and placebo at Day 4
The difference in change of quality of life from baseline between D-mannose and placebo | Day 1 to 2
  The difference in change of quality of life from baseline between D-mannose and placebo assessed by the RAND SF-36 questionnaire at Day 2
The difference in change of quality of life from baseline between D-mannose and placebo | Day 1 to 3
  The difference in change of quality of life from baseline between D-mannose and placebo assessed by the RAND SF-36 questionnaire at Day 3
The difference in change of quality of life from baseline between D-mannose and placebo | Day 1 to 4
  The difference in change of quality of life from baseline between D-mannose and placebo assessed by the RAND SF-36 questionnaire at Day 4
The difference in proportion of participants taking rescue medication up to Day 4 and/or during the follow-up period between D-mannose and placebo | Day 1 to 7

OTHER OUTCOMES:
Incidence of pre-emergent and post-emergent adverse events (AE) | Day 1 to 7
Incidence of clinically relevant changes in blood pressure (BP) | Day 1 to 4
Incidence of clinically relevant changes in heart rate (HR) | Day 1 to 4
Incidence of clinically relevant changes in clinical chemistry | Day 1 to 4
  Incidence of clinically relevant changes in clinical chemistry (aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase (ALP), total bilirubin, creatinine, electrolytes (Na, K, Cl), and estimated glomerular filtration rate (eGFR)
Incidence of clinically relevant changes in hematology | Day 1 to 4
  Incidence of clinically relevant changes in hematology (white blood cell (WBC) count with differential (neutrophils, lymphocytes, monocytes, eosinophils, basophils), red blood cell (RBC) count, hemoglobin, hematocrit, platelet count, immature granulocytes, nucleated RBC, RBC indices (mean corpuscular volume (MCV), mean corpuscular hemoglobin (MCH), mean corpuscular hemoglobin concentration (MCHC), red cell distribution width (RDW)

CONTACTS AND LOCATIONS:
Overall Officials: David Crowley, MD, Principal Investigator — KGK Science Inc.
Locations (1):
- KGK Science Inc., London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No